CLINICAL TRIAL: NCT01056341
Title: A Randomised, Controlled, Multidose, Multicentre, Adaptive Phase II/III Study in Infants With Proliferating Infantile Hemangiomas (IHs) Requiring Systemic Therapy to Compare 4 Regimens of Propranolol (1 or 3 mg/kg/Day for 3 or 6 Months) to Placebo (Double Blind).
Brief Title: Study to Demonstrate the Efficacy and Safety of Propranolol Oral Solution in Infants With Proliferating Infantile Hemangiomas Requiring Systemic Therapy
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Pierre Fabre Dermatology (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: V00400 SB 201 Study
Record Dates: First submitted 2010-01-24; First posted 2010-01-26 (Estimated); Results first posted 2014-06-24 (Estimated); Last update posted 2015-12-10 (Estimated); Status verified 2015-11

CONDITIONS: Infantile Hemangioma
Keywords: Infantile Hemangioma; Propranolol
MeSH Terms: conditions — Hemangioma, Capillary | interventions — Propranolol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Propranolol oral solution (Experimental)
  Interventions: Drug: Propranolol
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Propranolol — Propranolol (1 or 3 mg/kg/day for 3 or 6 months)
  Arms: Propranolol oral solution
Drug: Placebo — Treatment with placebo for 6 months
  Arms: Placebo

SUMMARY:
There is an unsatisfied medical need for a first-line treatment of proliferating IHs with a good benefit/risk profile. Based on the recent findings of encouraging results obtained with propranolol in a series of infants with severe Infantile Hemangioma (IH), propranolol is expected to be of significant benefit in the management of the condition. The present study has been designed to confirm efficacy of propranolol in severe IH by demonstrating superiority over placebo and to document the safety profile of propranolol in this indication.

DETAILED DESCRIPTION:
Primary objective The primary objective of this study is to identify the appropriate dose and duration of propranolol treatment and demonstrate its superiority over placebo based on the complete/nearly complete resolution of target IH at W24.

ELIGIBILITY:
Inclusion Criteria:

* Proliferating IH (target hemangioma) requiring systemic therapy anywhere on the body except on the diaper area with largest diameter of at least 1.5 cm

Exclusion Criteria:

- The patient presents with one or more of the following medical conditions: Congenital hemangioma; Kasabach-Merritt syndrome; bronchial asthma; bronchospasm; hypoglycaemia (< 40 mg/dl or at risk); untreated phaeochromocytoma; hypotension (< 50/30 mmHg); second or third degree heart block; cardiogenic shock; metabolic acidosis; bradycardia (< 80 bpm); severe peripheral arterial circulatory disturbances; Raynaud's phenomenon; sick sinus syndrome; uncontrolled heart failure or Prinzmetal's angina; documented PHACES syndrome with central nervous system involvement

* The patient has previously been treated for IH, including any surgical and/or medical procedures (e.g. laser therapy)
* The patient is known to have a hypersensitivity to propranolol and/or any other beta-blockers
* One or more of the following types of IH are present:

  * Life-threatening IH
  * Function-threatening IH (e.g. those causing impairment of vision, respiratory compromise caused by airway lesions, etc.)
  * Ulcerated IH (whatever the localisation) with pain and lack of response to simple wound care measures
* The patient was born prematurely and has not yet reached his/her term equivalent age (e.g. an infant born 2 months prematurely cannot be included before the age of 2 months)
* LVEF (left ventricular systolic function) ≤40% and/or cardiomyopathy and/or hereditary arrhythmia disorder

Ages: 35 Days to 150 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 512 (Actual)
Dates: Start 2010-01; Primary Completion 2012-05 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christine Labreze, MD, Study Chair — Hopital de Bordeaux
Locations (59):
- United States (10):
  - University of California, Irvine, California
  - Lucile Packard Children's Hospital, Redwood City, California
  - Rady Children's Hospital, San Diego, California
  - Miami Children's Hospital, Miami, Florida
  - Children's Memorial Hospital, Chicago, Illinois
  - Cardinal Glennon Children's Hospital, St Louis, Missouri
  - State University of NY, Brooklyn, New York
  - Oregon Health Sciences University, Portland, Oregon
  - Dell Children's Medical center, Austin, Texas
  - Seattle Children's Hospital, Seattle, Washington
- Australia (3):
  - Eastern Clinical Research Unit - Box Hill Hospital, Box Hill
  - Royal Children's Hospital, Melbourne
  - Sydney Children's Hospital, Randwick
- Canada (2):
  - CHU St.Justine, Montreal
  - The Hospital for Sick Children, Toronto
- Czechia (2):
  - Children Dermatology, Brno
  - Clinic of Dermatovenerology, University, Prague
- France (10):
  - Hôpital Pellegrin-Enfants, Bordeaux
  - Hôpital Femme Mère Enfant, Lyon
  - CHU Hôtel Dieu, Nantes
  - Hôpital Archet 2, Nice
  - Hôpital Armand Trousseau, Paris
  - Hôpital Necker Enfants malades, Paris
  - Hopital Robert Debre - Consultation de Dermatologie, Paris
  - Hopital Nord-CHU St Etienne, Saint-Etienne
  - Hôpital des enfants, Toulouse
  - Hôpital Clocheville, Tours
- Germany (4):
  - Universitätsklinikum Freiburg, Freiburg im Breisgau
  - Kinderkrankenhaus Wilhelmstift, Hamburg
  - Universitätsklinikum Schleswig-Holstein, Kiel
  - Kinderchirurgische Klinik Ludwig-Maximilians-Universität, München
- Heim Pál Gyermekkórház,, Budapest, Hungary
- Italy (2):
  - University of Bari, Bari
  - Clinica Dermatologica, Milan
- Vilnius University Children's Hospital, Vilnius, Lithuania
- Hospital Infantil de Mexico Federico Gomez, Mexico City, Mexico
- New Zealand (2):
  - Auckland Dermatology, Auckland
  - Waikato Clinical Research 2008 Ltd., Hamilton
- Peru (3):
  - Clinica Internacional, Lima
  - Hospital Nacional Edgardo Rebagliati Martins, Lima
  - Instituto Nacional de Salud del Niño, Lima
- Poland (4):
  - Klinika Chirurgii i Urologii Dzieci i Mlodziezy Akademii Medycznej, Gdansk
  - University Children's Hospital, Krakow
  - Department of Pediatric Surgery and Oncology, Lodz
  - Klinika Onkologii, Centrum Zdrowia Dziecka, Warsaw
- Romania (5):
  - Spitalul Clinic Urgenta pentru Copii Grigore Alexandrescu, Bucharest
  - I.O.M.C Alfred Rusescu, Bucharest
  - Spitalul de Copii Dr. Victor Gomoiu, Bucharest
  - Spitalul Clinic de Urgenta pentu Copii Sf. Maria, Iași
  - Spitalul de Urgenta Copii, Louis Turcanu, Timișoara
- Russia (3):
  - Medical University - Filatov Pediatric Hospital, Moscow
  - Medical Pediatric Academy, St-Peterburg
  - Neonatal Intensive Care Department, St-Peterburg
- Spain (6):
  - Servicio de Dermatologia del Hospital Infantil, A Coruña
  - Hospital Sant Pau de Barcelona, Barcelona
  - Hospital Universitario Infantil Niño Jesús, Madrid
  - Hospital La Paz, Madrid
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Universitario de Valencia, Valencia

REFERENCES:
- [Background] Leaute-Labreze C, Dumas de la Roque E, Hubiche T, Boralevi F, Thambo JB, Taieb A. Propranolol for severe hemangiomas of infancy. N Engl J Med. 2008 Jun 12;358(24):2649-51. doi: 10.1056/NEJMc0708819. No abstract available. PMID 18550886
- [Background] Sans V, de la Roque ED, Berge J, Grenier N, Boralevi F, Mazereeuw-Hautier J, Lipsker D, Dupuis E, Ezzedine K, Vergnes P, Taieb A, Leaute-Labreze C. Propranolol for severe infantile hemangiomas: follow-up report. Pediatrics. 2009 Sep;124(3):e423-31. doi: 10.1542/peds.2008-3458. Epub 2009 Aug 10. PMID 19706583
- [Result] Leaute-Labreze C, Hoeger P, Mazereeuw-Hautier J, Guibaud L, Baselga E, Posiunas G, Phillips RJ, Caceres H, Lopez Gutierrez JC, Ballona R, Friedlander SF, Powell J, Perek D, Metz B, Barbarot S, Maruani A, Szalai ZZ, Krol A, Boccara O, Foelster-Holst R, Febrer Bosch MI, Su J, Buckova H, Torrelo A, Cambazard F, Grantzow R, Wargon O, Wyrzykowski D, Roessler J, Bernabeu-Wittel J, Valencia AM, Przewratil P, Glick S, Pope E, Birchall N, Benjamin L, Mancini AJ, Vabres P, Souteyrand P, Frieden IJ, Berul CI, Mehta CR, Prey S, Boralevi F, Morgan CC, Heritier S, Delarue A, Voisard JJ. A randomized, controlled trial of oral propranolol in infantile hemangioma. N Engl J Med. 2015 Feb 19;372(8):735-46. doi: 10.1056/NEJMoa1404710. PMID 25693013

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 512 patients were included in the study (informed Consent Form signed). Among these 510 patients, 460 were randomized and 52 were screen failure
  * At least one inclusion criterion not met in 26 cases
  * Parent's decision in 12 cases
  * Other reasons in 15 cases.
  One patient was not included for two reasons (Parent's decision and other reason)
Groups:
- Propranolol 1mg/kg/d 3 Months: Propranolol oral solution 1mg/kg/day for 3 months, then placebo for 3 months
- Propranolol 1 mg/kg/d 6 Months: Propranolol oral solution 1mg/kg/day for 6 months
- Propranolol 3 mg/kg/d 3 Months: Propranolol oral solution 3mg/kg/day for 3 months, then placebo for 3 months
- Propranolol 3 mg/kg/d 6 Months: Propranolol oral solution 3mg/kg/day for 6 months
Period: Overall Study
Arm/Group | Placebo | Propranolol 1mg/kg/d 3 Months | Propranolol 1 mg/kg/d 6 Months | Propranolol 3 mg/kg/d 3 Months | Propranolol 3 mg/kg/d 6 Months
Started | 55 | 99 | 103 | 101 | 102
Interim Analysis | 25 | 41 | 41 | 40 | 43
Completed | 19 | 63 | 88 | 65 | 88
Not Completed | 36 | 36 | 15 | 36 | 14
Not completed — Treatment Intolerance | 0 | 2 | 0 | 2 | 0
Not completed — Lack of Efficacy | 32 | 30 | 7 | 25 | 9
Not completed — Other reasons | 4 | 4 | 8 | 9 | 5

BASELINE CHARACTERISTICS:
Population: Among the 460 randomized patients, 4 were not treated: 2 because of parent(s)'/guardian's decision (1 in 1mg/kg/day 6 months arm,1 in 3 mg/kg/day 3 months arm), 2 because of absence of adequate treatment on site (1 in 1 mg/kg/day 3 months arm and 1 in 3mg/kg/day 6 months arm).
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Propranolol 1mg/kg/d 3 Months | Propranolol 1 mg/kg/d 6 Months | Propranolol 3 mg/kg/d 3 Months | Propranolol 3 mg/kg/d 6 Months | Total
Number analyzed (Participants) | 55 | 98 | 102 | 100 | 101 | 456
Age, Continuous [Mean (Standard Deviation); unit: DAYS] | 103.91 (31.06) | 103.58 (33.07) | 102.65 (30.12) | 107.53 (30.14) | 101.63 (31.00) | 103.85 (31.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 68 | 70 | 79 | 70 | 325
  Male | 17 | 30 | 32 | 21 | 31 | 131
Region of Enrollment [Number; unit: participants]
  United States | 6 | 13 | 13 | 11 | 10 | 53
  Spain | 5 | 9 | 14 | 17 | 14 | 59
  Lithuania | 1 | 7 | 4 | 1 | 5 | 18
  Russian Federation | 0 | 1 | 0 | 1 | 1 | 3
  Italy | 1 | 0 | 0 | 0 | 1 | 2
  France | 21 | 25 | 18 | 22 | 28 | 114
  Czech Republic | 2 | 1 | 3 | 1 | 1 | 8
  Hungary | 1 | 2 | 4 | 2 | 2 | 11
  Mexico | 0 | 2 | 0 | 3 | 0 | 5
  Canada | 2 | 5 | 6 | 3 | 2 | 18
  Poland | 4 | 4 | 6 | 8 | 4 | 26
  Romania | 2 | 2 | 1 | 0 | 2 | 7
  Peru | 1 | 5 | 9 | 8 | 12 | 35
  Australia | 1 | 5 | 14 | 5 | 7 | 32
  Germany | 8 | 17 | 9 | 17 | 9 | 60
  New Zealand | 0 | 0 | 1 | 1 | 3 | 5
Infantile hemangioma localization [Number; unit: participants]
  FACE | 40 | 71 | 72 | 64 | 71 | 318
  NONE FACE | 15 | 27 | 30 | 36 | 30 | 138

OUTCOME MEASURES:

1. Primary Outcome: Interim Analysis : Complete/Nearly Complete Resolution of the Target Infantile Hemangioma at Week 24 Compared to Baseline Based on the Intra-patient Blinded Centralized Independent Qualitative Assessments of Week 24 Photographs.
Time Frame: 6 months
Population: Among the 190 first randomized patients who entered the stage 1 of the study, 2 patients were not treated because of parent'/legal guardian's decision: 1 in the 1mg/kg/day 6 months arm and 1 in the 3 mg/kg/day 3 months arm.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Propranolol 1mg/kg/d 3 Months | Propranolol 1 mg/kg/d 6 Months | Propranolol 3 mg/kg/d 3 Months | Propranolol 3 mg/kg/d 6 Months
Number analyzed (Participants) | 25 | 41 | 40 | 39 | 43
percentage of participants | 8.0 | 9.8 | 37.5 | 7.7 | 62.8
Statistical Analysis 1: Comparison: Placebo vs Propranolol 1mg/kg/d 3 Months vs Propranolol 1 mg/kg/d 6 Months vs Propranolol 3 mg/kg/d 3 Months vs Propranolol 3 mg/kg/d 6 Months; The interim analysis was carried out after the first 188 patients have completed their W24 visit or been withdrawn prematurely from study therapy. For each propranolol arm, individual hypotheses H0,i: θi≤0; Test type: Superiority or Other; p < 0.0001, One-sided Z-tests — P-value not adjusted for multiplicity. An Independent Committee conducted this analysis to determine the most efficacious of all arms with a good safety profile. P-value linked to the 3 mg/kg/day 6 months selected arm; One-sided Z-tests for proportions (contrasts tests on placebo) with pooled variance

2. Primary Outcome: Primary Analysis : Complete/Nearly Complete Resolution of the Target Infantile Hemangioma at W24 Compared to Baseline Based on the Intra-patient Blinded Centralized Independent Qualitative Assessments of W24 Photographs.
Time Frame: 6 months
Population: After the interim analysis results, the Independent Committee recommendations was to continue the trial with the 3 mg/kg/day6 months arm and the placebo arm. 55 randomized and treated patients in the placebo arm and 102 randomized patients in the 3 mg/kg/day6 months arm,1 was not treated because no unit of the assigned treatment available on site.
Measure: Number; unit: percentage of participants
Groups:
- Propranolol 3mg/kg/d 6 Months: Propranolol 3 mg/kg/day for 6 months
Arm/Group | Placebo | Propranolol 3mg/kg/d 6 Months
Number analyzed (Participants) | 55 | 101
percentage of participants | 3.6 | 60.4
Statistical Analysis 1: Comparison: Placebo vs Propranolol 3mg/kg/d 6 Months; The objective is to test the superiority of the selected arm using the approach of Posch et al. The primary analysis was performed on the intent-to-treat population: all treated patients in Stage 1 and all treated patients in stage 2 randomized to placebo or the selected arm; Test type: Superiority or Other; p < 0.0001, combination tests — The methodology used guaranteed that the familywise type I error rate was below the nominal one-sided significance level of 0.005; Superiority was tested using the closed testing procedure and combination tests for all intersection hypotheses using Simes' adjustment

3. Secondary Outcome: Success/Failure Based on the Investigator Qualitative Assessment of Complete Resolution at W48.
Description: Time to first sustained improvement based on centralized qualitative assessments of paired patient-visits
Time Frame: 6 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Safety evaluation of the four regimens of oral propranolol (versus placebo) over a 24-week treatment period. Safety evaluation of the four previous regimens of oral propranolol (versus placebo) over a follow up period of 72 weeks (up to 96 weeks).
Description: Safety population included all participants who received at least one dose of Propranolol (1 or 3mg/kg/day for 3 or 6 months) or placebo.
  Among the 456 treated patients, 65 were withdrawn during treatment period:22 in placebo arm, 13 in 1mg/kg/day 3months arm, 11 in 1mg/kg/day 6months arm, 13 in 3mg/kg/day 3months arm, 6 in 3mg/kg/day 6months arm.
Groups:
- W24-treatment Period-safety Set-Placebo: Placebo: Treatment with placebo for 6 months
- W24-treatment Period-safety Set-Propranolol 1mg/kg/d 3 Months: Propranolol hydrochloride oral solution 1mg/kg/day for 3 months, then placebo for 3 months
- W24-treatment Period-safety Set-Propranolol 1 mg/kg/d 6 Months: Propranolol hydrochloride oral solution 1mg/kg/day for 6 months
- W24-treatment Period-safety Set-Propranolol 3 mg/kg/d 3 Months: Propranolol hydrochloride oral solution 3mg/kg/day for 3 months, then placebo for 3 months
- W24-treatment Period-safety Set-Propranolol 3 mg/kg/d 6 Months: Propranolol hydrochloride oral solution 3mg/kg/day for 6 months
- W72-follow-up Period of ex Placebo Group-safety Set; W72-follow-up Period of ex 1mg/kg/d 3 Months Group-safety Set; W72-follow-up Period of ex 1mg/kg/d 6 Months Group-safety Set; W72-follow-up Period of ex 3mg/kg/d 3 Months Group-safety Set; W72-follow-up Period of ex 3mg/kg/d 6 Months Group-safety Set: 72-week follow-up period without study treatment administration
Arm/Group | W24-treatment Period-safety Set-Placebo | W24-treatment Period-safety Set-Propranolol 1mg/kg/d 3 Months | W24-treatment Period-safety Set-Propranolol 1 mg/kg/d 6 Months | W24-treatment Period-safety Set-Propranolol 3 mg/kg/d 3 Months | W24-treatment Period-safety Set-Propranolol 3 mg/kg/d 6 Months | W72-follow-up Period of ex Placebo Group-safety Set | W72-follow-up Period of ex 1mg/kg/d 3 Months Group-safety Set | W72-follow-up Period of ex 1mg/kg/d 6 Months Group-safety Set | W72-follow-up Period of ex 3mg/kg/d 3 Months Group-safety Set | W72-follow-up Period of ex 3mg/kg/d 6 Months Group-safety Set
Serious Adverse Events (participants affected / at risk) | 3/55 | 5/98 | 3/102 | 9/100 | 5/101 | 5/33 | 6/85 | 5/91 | 5/87 | 7/95
Other Adverse Events (participants affected / at risk) | 40/55 | 88/98 | 92/102 | 92/100 | 96/101 | 27/33 | 66/85 | 70/91 | 65/87 | 75/95
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | W24-treatment Period-safety Set-Placebo (N=55) | W24-treatment Period-safety Set-Propranolol 1mg/kg/d 3 Months (N=98) | W24-treatment Period-safety Set-Propranolol 1 mg/kg/d 6 Months (N=102) | W24-treatment Period-safety Set-Propranolol 3 mg/kg/d 3 Months (N=100) | W24-treatment Period-safety Set-Propranolol 3 mg/kg/d 6 Months (N=101) | W72-follow-up Period of ex Placebo Group-safety Set (N=33) | W72-follow-up Period of ex 1mg/kg/d 3 Months Group-safety Set (N=85) | W72-follow-up Period of ex 1mg/kg/d 6 Months Group-safety Set (N=91) | W72-follow-up Period of ex 3mg/kg/d 3 Months Group-safety Set (N=87) | W72-follow-up Period of ex 3mg/kg/d 6 Months Group-safety Set (N=95)
Apathy (Psychiatric disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Atrioventricular block second degree (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bronchiolitis (Infections and infestations) | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 2
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 0
Bronchopneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Condition aggravated (General disorders) | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cyanosis (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cystitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Drug ineffective (General disorders) | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Enterocolitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Epilepsy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Traumatic brain injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ileostomy closure (Surgical and medical procedures) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Inguinal hernia repair (Surgical and medical procedures) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rotavirus infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 2 | 0
Viraemia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
cataract operation (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
surgery (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Finger amputation (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
hip surgery (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
hospitalisation (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
scrotal operation (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
hip dysplasia (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
asphyxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
convulsion (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
febrile convulsion (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
inflammation (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
hyperthermia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
ketoacidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
type 1 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
respiratory tract infection viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
ear infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
gastroenteritis rotavirus (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
otitis media acute (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
respiratory syncytial virus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
tonsillitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | W24-treatment Period-safety Set-Placebo (N=55) | W24-treatment Period-safety Set-Propranolol 1mg/kg/d 3 Months (N=98) | W24-treatment Period-safety Set-Propranolol 1 mg/kg/d 6 Months (N=102) | W24-treatment Period-safety Set-Propranolol 3 mg/kg/d 3 Months (N=100) | W24-treatment Period-safety Set-Propranolol 3 mg/kg/d 6 Months (N=101) | W72-follow-up Period of ex Placebo Group-safety Set (N=33) | W72-follow-up Period of ex 1mg/kg/d 3 Months Group-safety Set (N=85) | W72-follow-up Period of ex 1mg/kg/d 6 Months Group-safety Set (N=91) | W72-follow-up Period of ex 3mg/kg/d 3 Months Group-safety Set (N=87) | W72-follow-up Period of ex 3mg/kg/d 6 Months Group-safety Set (N=95)
Bronchiolitis (Infections and infestations) | 3 | 5 | 7 | 5 | 9 | 2 | 6 | 4 | 9 | 11
Bronchitis (Infections and infestations) | 1 | 5 | 8 | 10 | 16 | 3 | 12 | 14 | 18 | 20
Conjunctivitis (Eye disorders) | 2 | 4 | 8 | 2 | 8 | 1 | 7 | 8 | 7 | 9
Constipation (Gastrointestinal disorders) | 1 | 9 | 6 | 9 | 4 | 1 | 1 | 4 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 14 | 18 | 16 | 14 | 4 | 8 | 5 | 7 | 7
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 2 | 4 | 5 | 4 | 9 | 1 | 4 | 2 | 3 | 3
Diarrhea (Gastrointestinal disorders) | 4 | 16 | 14 | 17 | 28 (51) | 1 | 4 | 4 | 10 | 9
Ear infection (Infections and infestations) | 0 | 7 | 6 | 7 | 4 | 6 | 13 | 13 | 14 | 17
Eczema (Skin and subcutaneous tissue disorders) | 1 | 8 | 4 | 2 | 2 | 2 | 4 | 2 | 4 | 4
Gastroenteritis (Infections and infestations) | 2 | 2 | 5 | 4 | 11 | 4 | 7 | 9 | 14 | 14
Insomnia (Psychiatric disorders) | 3 | 3 | 1 | 3 | 3 | 1 | 0 | 0 | 0 | 0
Irritability (General disorders) | 3 | 5 | 6 | 1 | 2 | 0 | 0 | 1 | 0 | 0
Middle insomnia (Psychiatric disorders) | 3 | 6 | 4 | 7 | 6 | 0 | 0 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 10 | 29 | 21 | 32 | 34 | 8 | 26 | 20 | 24 | 30
Peripheral coldness (Vascular disorders) | 1 | 8 | 10 | 1 | 10 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 6 | 21 | 24 | 22 | 28 | 6 | 21 | 15 | 20 | 24
Rhinitis (Infections and infestations) | 5 | 13 | 13 | 5 | 5 | 3 | 9 | 7 | 1 | 6
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 3 | 8 | 3 | 0 | 0 | 0 | 3 | 5
Sleep disorder (Psychiatric disorders) | 1 | 12 | 6 | 1 | 7 | 1 | 1 | 0 | 1 | 1
Somnolence (Nervous system disorders) | 1 | 6 | 4 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Teething (Gastrointestinal disorders) | 6 | 19 | 23 | 16 | 22 | 0 | 5 | 9 | 7 | 8
Toothhache (Gastrointestinal disorders) | 2 | 5 | 2 | 8 | 10 | 0 | 1 | 0 | 0 | 4
Upper respiratory tract infection (Infections and infestations) | 4 | 6 | 13 | 20 | 16 | 5 | 7 | 15 | 13 | 11
Vaccination complication (Injury, poisoning and procedural complications) | 2 | 7 | 9 | 8 | 8 | 1 | 1 | 1 | 2 | 2
Vomiting (Gastrointestinal disorders) | 3 | 16 | 13 | 10 | 13 | 2 | 3 | 3 | 4 | 2
nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 6 | 4 | 4 | 0 | 1 | 1 | 0 | 1
asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 2 | 0 | 2 | 3 | 5 | 5
hypotonia (Nervous system disorders) | 0 | 1 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0
condition aggravated (General disorders) | 0 | 3 | 1 | 3 | 2 | 2 | 1 | 1 | 1 | 3
agitation (Psychiatric disorders) | 0 | 1 | 6 | 3 | 0 | 0 | 0 | 0 | 0 | 0
gingival pain (Gastrointestinal disorders) | 1 | 3 | 0 | 5 | 2 | 1 | 1 | 0 | 1 | 0
dermatitis atopic (Skin and subcutaneous tissue disorders) | 1 | 2 | 1 | 1 | 3 | 2 | 0 | 0 | 2 | 2
decreased appetite (Metabolism and nutrition disorders) | 1 | 5 | 3 | 5 | 1 | 0 | 0 | 1 | 0 | 1
tonsillitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 3 | 7 | 6 | 7 | 10
pharyngitis (Infections and infestations) | 0 | 4 | 3 | 2 | 3 | 0 | 5 | 4 | 6 | 8
otite media (Infections and infestations) | 0 | 1 | 1 | 3 | 2 | 6 | 5 | 4 | 4 | 5
influenza (Infections and infestations) | 1 | 1 | 3 | 3 | 4 | 1 | 2 | 0 | 2 | 5
varicella (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 5 | 4 | 6 | 4
roseola (Infections and infestations) | 1 | 1 | 0 | 2 | 0 | 1 | 3 | 5 | 1 | 4
hand-foot-and-mouth disease (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 2 | 3 | 3
acute tonsillitis (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 2 | 1 | 0 | 1 | 2
croup infectious (Infections and infestations) | 0 | 1 | 1 | 0 | 1 | 2 | 1 | 1 | 1 | 1
eye infection (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 3 | 0 | 0 | 1 | 0
gastroenteritis viral (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigators can reserve the right to publish or present study data; provided that the sponsor reviews the abstract or manuscript at least 60 days prior to the expected date of submission to the intended publisher or planned presentation.

Publication of study results by each site shall be made only after completion and finalisation of the study by all sites and first publication by the Sponsor.